CLINICAL TRIAL: NCT01093963
Title: Adjunctive Lisdexamfetamine in Bipolar Depression
Brief Title: Efficacy Study of Lisdexamfetamine to Treat Bipolar Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment goals not met
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Shire (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDX BP
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine (Active Comparator): Drug
  Interventions: Drug: Lisdexamfetamine
- Placebo (Placebo Comparator): Drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine — oral; 20-70mg/day
  Arms: Lisdexamfetamine
Drug: Placebo — oral; 20-70mg/day
  Arms: Placebo

SUMMARY:
The specific aim of this study is to evaluate the efficacy and tolerability of a stimulant (lisdexamfetamine) in the adjunctive treatment of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, through the ages of 18 and 55 years, inclusive.

Exclusion Criteria:

* Women who are pregnant, lactating, or of childbearing potential who are not using adequate contraceptive measures.
* Subjects who are displaying clinically significant homicidality or suicidality
* Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease. Subjects should be biochemically euthyroid to enter the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in the Montgomery-Asberg Depression Rating Scale | 30-36 months
  Efficacy will be assessed by measuring the baseline-to-endpoint change in the Montgomery-Asberg Depression Rating Scale (MADRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Lindner Center of HOP, Mason, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Martens BE, Mori N, Blom TJ, Casuto LS, Hawkins JM, Keck PE Jr. Adjunctive lisdexamfetamine in bipolar depression: a preliminary randomized, placebo-controlled trial. Int Clin Psychopharmacol. 2015 Jan;30(1):6-13. doi: 10.1097/YIC.0000000000000051. PMID 25340384